CLINICAL TRIAL: NCT06515704
Title: The Mental Health of Young Adults in Times of Polycrisis
Brief Title: Mental Health of the Polycrisis Generation
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Bernadetta Izydorczyk, Prof. dr hab., Jagiellonian University
Other Study IDs: Polycrisis
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-08

CONDITIONS: Stress; Stress-related Problem; Cumulative Trauma; Mental Health Issue; Mental Stress; Quality of Life
Keywords: cumulative stress; quality of life; mental health; young adults; stress syndrome; resilience; closeness relationships; postformal thinking; personality; development; risk factors; protective factors
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- A representative sample of Polish young adults: Polish young adults, aged 18-29, living in Poland during this period (2020-2023:
  COVID-19, lockdown, economic crisis, political changes, climate changes, and the war in Ukraine). Intervention: psychological tests and psychosocial questionnaires Assessment of psychological functioning (including quality of life, mental health conditions, coping skills- adaptation to stress, global crisises, developmental crisis; resilience; postformal thinking; relationships with parents/ partners/ friends), and socio-demographics, academic performance, home, general health, habits, and attitudes.

SUMMARY:
The goal of this observational, longitudinal study is to identify risk and protective factors that buffer the effects of individual daily stress and adaptation to global crises on the quality of life and mental health conditions of young people entering adulthood (aged 18-29, fluent in Polish, and living in Poland). Moderators such as factors related to development, personality variables compatible with the domains according to ICD-11, psychological resilience, closeness in relationships with a partner/friends/parents, and the level of postformal thinking will also be considered.

The main hypotheses it aims to consider are:

H1: Poorer adaptation to individual and global crises is associated with higher levels of perceived stress, leading to worse indicators of mental health and quality of life.

H2: A higher level of implementation of developmental tasks, including more fulfilled criteria of adulthood and a mature identity, mitigates the relationship between stress/ crisis adaptation and health and quality of life indicators.

H3: Resilience and better relationships (closeness with a partner/ friends/ parents) buffer the negative effect of stress on health and quality of life.

H4: A higher level of postformal thinking mitigates the relationship between stress/ crisis adaptation and health and quality of life indicators.

H5: A higher intensity of psychopathological personality traits is a risk factor that amplifies the negative effect of stress on health and quality of life.

Researchers will analyze measurements taken from the same group (a representative sample of Polish young adults) at two time points - now and in 12 months. The aim is to observe the extent to which the effects of current daily stressors and adaptation to the crisis, as well as the effects of potential moderators, are relatively stable.

DETAILED DESCRIPTION:
Background: The WHO and other international organizations clearly indicate the co-occurrence of multiple health problems and an increasing trend in the deterioration of mental health among young people. This is related to the experience of cumulative stress, generally referred to as a 'polycrisis', which involves the simultaneous occurrence of crises such as the COVID-19 pandemic, displacements and trauma resulting from the war in Ukraine, and climate change.

An additional factor is the stress of daily life and everyday challenges. These latter seem particularly important during the period when an individual faces some of the greatest challenges, such as entering young adulthood and taking on adult roles. However, there is a lack of studies analyzing the risk factors and protective factors that buffer the impact of contemporary cumulative stress on the mental health of young adults in different cultures (including Polish).

Participants: a representative population of 600 Polish young adults, aged 18-29.

Methodology: Analysis of data collected through psychological scales and questionnaires related to daily stress, adaptation to global crises, mental health conditions, quality of life, meeting mature developmental criteria, personality traits, resilience, closeness in relationships, and postformal thinking.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 29 years
* Standard educational opportunities
* Polish fluent
* Polish nationality

Exclusion Criteria:

* Intellectual disability
* Inability to self-complete the research questionnaires

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults, Polish representative sample, aged 18-29
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The International Adjustment Disorder Questionnaire (IADQ) | September 01, 2024 until September 30, 2024
  Polish version of IADQ is a brief, simply-worded measure, focusing only on the core features of Adjustment Disorder, and employs straightforward diagnostic rules. The IADQ was developed to be consistent with the organizing principles of the ICD-11, as set forth by the World Health Organization, which are to maximize clinical utility and ensure international applicability through a focus on the core symptoms of a given disorder. A probable diagnosis of Adjustment Disorder requires the presence of (1) a psychosocial stressor (score ≥ 1 on the IADQ stressor list, items 1-9), (2) at least one 'Preoccupation' symptom (items 10- 12) rated ≥ 2), (3) at least one 'Failure to Adapt' symptom (items 13-15) rated ≥ 2, (4) symptoms began within one month of the stressor (positive endorsement of item 16), and (5) evidence of functional impairment indicated by any of item 17-19 rated ≥ 2).
The International Adjustment Disorder Questionnaire (IADQ) - POLI | September 01, 2024 until September 30, 2024
  Polish, brief, simply-worded measure, based on IADQ, focusing on emotional adaptation to daily stress events. The calculation algorithm of IADQ is being developed by the research team (standardization).
Perceived Stress Scale (PPS-10) | September 01, 2024 until September 30, 2024
  The PSS-10 is used to measure perceived stress. It contains 10 questions related to various subjective feelings associated with personal problems and events, behaviors, and coping methods. It is used to assess the intensity of stress related to one's life situation over the past month. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 27-40 would be considered high perceived stress.
Personality Traits (PiCD) | September 01, 2024 until September 30, 2024
  Personality Inventory for ICD-11 (PiCD). The four-factor structure of the Polish version of PiCD consists of three unipolar factors as Negative Affectivity, Detachment, and Dissociality factors, and one bipolar Anankastia vs. Disinhibition factor. According to Polish standardization, symptom severity is indicated by scores above one standard deviation from the mean.
The Dimensions of Identity Development Scale (DIDS) | September 01, 2024 until September 30, 2024
  The DIDS is a scale measuring identity processes in five domains: exploration in breadth, commitment making, exploration in depth, identification with commitment, and ruminative exploration. Each of the five dimensions is measured by 5 items, assessed on a 5-point Likert scale. According to Polish standardization, symptom severity is indicated by scores above one standard deviation from the mean.
The Markers of Adulthood | September 01, 2024 until September 30, 2024
  The scale for assessing the fulfillment of adulthood criteria according to Nelson and Barry in the areas of: independence, interdependence, role transitions, conformity to norms, biological transitions, chronological transitions, family potential, and subjective perception of adulthood. The scale is qualitative in nature. Five dimensions of identity development:
  Exploration in breadth: Seeking alternatives for goals and values. Commitment making: Making choices and commitments. Exploration in depth: Evaluating commitments against personal standards. Identification with commitments: Confidence and internalization of choices. Ruminative exploration: Concerns and challenges in identity development, possibly indicating a crisis.
The Resilience Measure Questionnaire (KOP-26) | September 01, 2024 until September 30, 2024
  KOP-26, by Gąsior, Chodkiewicz and Cechowski, consists of 26 items referring to the protective factors linked with personal and social competences as well as family relations. Each of the three dimensions is measured by items assessed on a 5-point Likert scale. The higher the sum of points in a given area, the higher the competencies.
Closeness to biological mother and father questionnaire | September 01, 2024 until September 30, 2024
  The Polish adaptation of the Closeness to Biological Mother and Father Questionnaire consists of 6 questions regarding the relationship with the parent. Relationships with the mother and father are assessed separately each time on a 5-point scale.
Closeness to partner/ friend questionnaire | September 01, 2024 until September 30, 2024
  The Polish adaptation of the Closeness to Partner/Friend Questionnaire consists of 6 questions regarding the relationship with the partner. Relationships are assessed on a 5-point scale. The task of the respondent is to respond on a 5-point scale (1 means never, and 5 means always) to six questions concerning their relationship with the partner/friend. The task of the respondent is to respond on a 5-point scale (1 means never, and 5 means always) to six questions concerning their relationship with the partner/ friend.
Daily Problems Test | September 01, 2024 until September 30, 2024
  The Daily Problems Test by Gurba is based on the method of Sebby and Papini, who in the original version used the clinical method proposed, among others, by Piaget, based on asking questions such as "what?" and "why?". The test consists of three problems, which are translations of sample tasks by Sebby and Papini, relevant for adolescents, young adults, and aging adults.
The Mental Health Continuum-Short Form (MHC-SF) | September 01, 2024 until September 30, 2024
  The Polish adaptation of Mental Health Continuum-Short Form (MHC-SF) is the tool that allows for continuous assessment of subjective well-being (including its three aspects: emotional, psychological, and social), as well as for the categorical diagnosis of the presence of mental health and the absence of mental health (understood as flourishing and languishing). The answering scale is 6-points, and describes the frequency of experiencing various symptoms of well-being. The scale ranges from never to everyday (during the past month).
The World Health Organization Quality of Life (WHOQOL-PL) | September 01, 2024 until September 30, 2024
  The WHOQOL-PL is a Polish adaptation of the quality of life assessment developed by the WHOQOL Group, focusing on an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards, and concerns. The mean score of items within each domain is used to calculate the domain score. Domain scores are scaled in a positive directions (higher scores denote higher quality of life).
Authors survey | September 01, 2024 until September 30, 2024
  Survey of socio-demographic data (gender, age, sexual orientation, marital status, family, relationships, socioeconomic status, place of residence, educational level, habits, attitudes, others).

SECONDARY OUTCOMES:
The International Adjustment Disorder Questionnaire (IADQ) | September 30, 2025 until October 30, 2025
  Polish version of IADQ is a brief, simply-worded measure, focusing only on the core features of Adjustment Disorder, and employs straightforward diagnostic rules. The IADQ was developed to be consistent with the organizing principles of the ICD-11, as set forth by the World Health Organization, which are to maximize clinical utility and ensure international applicability through a focus on the core symptoms of a given disorder. A probable diagnosis of Adjustment Disorder requires the presence of (1) a psychosocial stressor (score ≥ 1 on the IADQ stressor list, items 1-9), (2) at least one 'Preoccupation' symptom (items 10- 12) rated ≥ 2), (3) at least one 'Failure to Adapt' symptom (items 13-15) rated ≥ 2, (4) symptoms began within one month of the stressor (positive endorsement of item 16), and (5) evidence of functional impairment indicated by any of item 17-19 rated ≥ 2).
The International Adjustment Disorder Questionnaire (IADQ) - POLI | September 30, 2025 until October 30, 2025
  Polish, brief, simply-worded measure, based on IADQ, focusing on emotional adaptation to daily stress events. The calculation algorithm of IADQ is being developed by the research team (standardization).
Perceived Stress Scale (PPS-10) | September 30, 2025 until October 30, 2025
  The PSS-10 is used to measure perceived stress. It contains 10 questions related to various subjective feelings associated with personal problems and events, behaviors, and coping methods. It is used to assess the intensity of stress related to one's life situation over the past month. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 27-40 would be considered high perceived stress.
Personality Traits (PiCD) | September 30, 2025 until October 30, 2025
  Personality Inventory for ICD-11 (PiCD). The four-factor structure of the Polish version of PiCD consists of three unipolar factors as Negative Affectivity, Detachment, and Dissociality factors, and one bipolar Anankastia vs. Disinhibition factor. According to Polish standardization, symptom severity is indicated by scores above one standard deviation from the mean.
The Dimensions of Identity Development Scale (DIDS) | September 30, 2025 until October 30, 2025
  The DIDS is a scale measuring identity processes in five domains: exploration in breadth, commitment making, exploration in depth, identification with commitment, and ruminative exploration. Each of the five dimensions is measured by 5 items, assessed on a 5-point Likert scale. According to Polish standardization, symptom severity is indicated by scores above one standard deviation from the mean.
The Markers of Adulthood | September 30, 2025 until October 30, 2025
  The scale for assessing the fulfillment of adulthood criteria according to Nelson and Barry in the areas of: independence, interdependence, role transitions, conformity to norms, biological transitions, chronological transitions, family potential, and subjective perception of adulthood. The scale is qualitative in nature. Five dimensions of identity development:
  Exploration in breadth: Seeking alternatives for goals and values. Commitment making: Making choices and commitments. Exploration in depth: Evaluating commitments against personal standards. Identification with commitments: Confidence and internalization of choices. Ruminative exploration: Concerns and challenges in identity development, possibly indicating a crisis.
The Resilience Measure Questionnaire (KOP-26) | September 30, 2025 until October 30, 2025
  KOP-26, by Gąsior, Chodkiewicz and Cechowski, consists of 26 items referring to the protective factors linked with personal and social competences as well as family relations. Each of the three dimensions is measured by items assessed on a 5-point Likert scale. The higher the sum of points in a given area, the higher the competencies.
Closeness to biological mother and father questionnaire | September 30, 2025 until October 30, 2025
  The Polish adaptation of the Closeness to Biological Mother and Father Questionnaire consists of 6 questions regarding the relationship with the parent. Relationships with the mother and father are assessed separately each time on a 5-point scale. The task of the respondent is to respond on a 5-point scale (1 means never, and 5 means always) to six questions concerning their relationship with the parent.
Closeness to partner/ friend questionnaire | September 30, 2025 until October 30, 2025
  The Polish adaptation of the Closeness to Partner/Friend Questionnaire consists of 6 questions regarding the relationship with the partner. Relationships are assessed on a 5-point scale. The task of the respondent is to respond on a 5-point scale (1 means never, and 5 means always) to six questions concerning their relationship with the partner/friend.
Daily Problems Test | September 30, 2025 until October 30, 2025
  The Daily Problems Test by Gurba is based on the method of Sebby and Papini, who in the original version used the clinical method proposed, among others, by Piaget, based on asking questions such as "what?" and "why?". The test consists of three problems, which are translations of sample tasks by Sebby and Papini, relevant for adolescents, young adults, and aging adults.
The Mental Health Continuum-Short Form (MHC-SF) | September 30, 2025 until October 30, 2025
  The Polish adaptation of Mental Health Continuum-Short Form (MHC-SF) is the tool that allows for continuous assessment of subjective well-being (including its three aspects: emotional, psychological, and social), as well as for the categorical diagnosis of the presence of mental health and the absence of mental health (understood as flourishing and languishing). The answering scale is 6-points, and describes the frequency of experiencing various symptoms of well-being. The scale ranges from never to everyday (during the past month). The mean score of items within each domain is used to calculate the domain score. Domain scores are scaled in a positive directions (higher scores denote higher quality of life).
The World Health Organization Quality of Life (WHOQOL-PL) | September 30, 2025 until October 30, 2025
  The WHOQOL-PL is a Polish adaptation of the quality of life assessment developed by the WHOQOL Group, focusing on an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards, and concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadetta Izydorczyk, Prof, Study Chair — Institute of Psychology, Jagiellonian University in Krakow, Poland; Anna Wendołowska, PhD, Principal Investigator — Institute of Psychology, Jagiellonian University in Krakow, Poland; Katarzyna Sitnik-Warchulska, PhD, Principal Investigator — Institute of Applied Psychology, Jagiellonian University in Krakow, Poland; Dorota Czyżowska, Prof., Principal Investigator — Institute of Psychology, Jagiellonian University in Krakow, Poland; Aleksandra Gruszka, Prof., Principal Investigator — Institute of Psychology, Jagiellonian University in Krakow, Poland; Weronika Kałwak, PhD, Principal Investigator — Institute of Psychology, Jagiellonian University in Krakow, Poland
Locations (2):
- Poland (2):
  - Behaviour in Crisis Lab, Impact of cumulative stress on the mental health of young people project, Jagiellonian University in Krakow, Krakow, Krakow
  - Behaviour in Crisis Lab, Jagiellonian University, Krakow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lawrance EL, Jennings N, Kioupi V, Thompson R, Diffey J, Vercammen A. Psychological responses, mental health, and sense of agency for the dual challenges of climate change and the COVID-19 pandemic in young people in the UK: an online survey study. Lancet Planet Health. 2022 Sep;6(9):e726-e738. doi: 10.1016/S2542-5196(22)00172-3. PMID 36087603
- [Background] Kauhanen L, Wan Mohd Yunus WMA, Lempinen L, Peltonen K, Gyllenberg D, Mishina K, Gilbert S, Bastola K, Brown JSL, Sourander A. A systematic review of the mental health changes of children and young people before and during the COVID-19 pandemic. Eur Child Adolesc Psychiatry. 2023 Jun;32(6):995-1013. doi: 10.1007/s00787-022-02060-0. Epub 2022 Aug 12. PMID 35962147
- [Background] Lloyd K, Schubotz D, Roche R, Manzi J, McKnight M. A Mental Health Pandemic? Assessing the Impact of COVID-19 on Young People's Mental Health. Int J Environ Res Public Health. 2023 Aug 9;20(16):6550. doi: 10.3390/ijerph20166550. PMID 37623136